CLINICAL TRIAL: NCT04075526
Title: Vancomycin Powder and Dilute Povidone Iodine Lavage for Infection Prophylaxis in High Risk Total Joint Arthroplasty
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-00851
Record Dates: First submitted 2019-08-29; First posted 2019-08-30 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Povidone-Iodine; Congresses as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Povidone iodine and vancomycin powder (Experimental)
  Interventions: Drug: Povidone iodine; Drug: Vancomycin powder
- Povidone iodine alone (Experimental)
  Interventions: Drug: Povidone iodine
- Vancomycin powder alone (Active Comparator)
  Interventions: Drug: Vancomycin powder
- Conventional (Active Comparator): neither povidone iodine, vancomycin powder, nor polymyxin/bacitracin irrigation
  Interventions: Other: Conventional

INTERVENTIONS:
Drug: Povidone iodine — To create the dilute solution, a staff member will draw up 17.5 mL of 10% povidone iodine with a syringe and mix it with 500 mL of normal saline, resulting in a dilution of 0.35% povidone iodine solution for use before wound closure.
  Arms: Povidone iodine alone; Povidone iodine and vancomycin powder
Drug: Vancomycin powder — 2 grams of vancomycin powder will be applied to the wound and will be distributed so that approximately 1 gram is administered deep to the fascia and 1 gram superficial to the fascia
  Arms: Povidone iodine and vancomycin powder; Vancomycin powder alone
Other: Conventional — No additional steps in management are required for the control arm of the study besides lavage with 1 L of isotonic sodium chloride solution without antibiotics. No vancomycin powder or dilute povidone iodine lavage would be utilized in this cohort
  Arms: Conventional

SUMMARY:
This is a prospective, randomized, controlled, open label, parallel four-arm design, multi-center study to compare different intraoperative interventions in the prevention of acute PJI development.

DETAILED DESCRIPTION:
The study seeks to define the potential benefits that an additional prophylactic protocol involving the use of povidone iodine and vancomycin powder on the incidence of PJI in high risk TJA patients. The potential benefits of these interventions are significant both from the perspective of reducing morbidity and mortality for the patient, and from a cost-effectiveness and value-based perspective. To this end, our study seeks to assess the direct and indirect costs associated with the treatment and control groups. We anticipate that the administration of a VPIP protocol will both reduce the incidence of PJI in high risk groups relative to the control arm and will demonstrate added value from a cost-effectiveness perspective.

This study looks to examine off-label use of Vancomycin Powder and Povidone Iodine 10% solution. Both products are lawfully marketed in the United States. This study is not intended to be reported to the FDA as a well-controlled study in support of a new indication and there is no intent to use it to support any other significant change in the labeling or advertising of either drug.

This study does not involve a route of administration, dose, patient population, or other factor that significantly increased the risk (or decreases the acceptability of the risk) associated with the use of the drug product. The routes and dosages being tested in this protocol are part of standard clinical care in most total joint arthroplasty surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Patient has no open wounds on operative leg
* Patient is scheduled to undergo elective primary and revision total joint arthroplasty for posttraumatic, osteoarthritis, avascular necrosis, and/or inflammatory arthritis
* Patient does not have active infection on the operative leg, the operative joint
* Patient are identified as high risk for the development of PJI which is determined by the presence of one or more of the following characteristics: BMI >35, active smoker, ASA ≥ 3, immunosuppressed (i.e. being treated with chemotherapy, diagnosis of HIV, diagnosis of HCV, being treated with chronic steroids, patients with inflammatory arthropathies), diagnosis with diabetes mellitus, established colonization with S. aureus, or any patient undergoing revision TJA
* Patient understand the risks and benefits associated with TJA and willing to cooperate and follow study protocol and visit schedule

Exclusion Criteria:

* Patient is pregnant
* Patient is unable to provide written consent
* Patient has psychiatric disorder that precludes safe study participation or that necessitates confinement in a custodial environment at home or in a chronic care facility
* Patient does not have the mental capacity to participate and comply with the study protocol
* Patient has active infections in the operative leg/joint
* Patient has severe dementia
* Suspicion of illicit drug abuse by patient
* ASA score of 5 & 6
* History of prior native septic joint arthritis
* No planned procedure within 90 days of surgery

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2129 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Rate of periprosthetic infection (PJI) after elective total joint arthroplasty. | 90 Days
  The definition of periprosthetic infection exists when the following criteria are met:
  * NEW MSIS criteria for PJI: 1 major criteria (2) or 6 minor criteria (6) 26-28
  * Major Criteria: [1] sinus tract [2] + Cx from 2 separate aspirations
  * Minor Criteria: [1] ESR >30 mm/hr (1 point), [2] D-dimer >860 ng/mL or CRP >1 mg/dL [2] increased synovial WBC (>3000 cells/microliter) [4] alpha-defensin (signal-to-cutoff ratio>1) [5] leukocyte esterase (++) [6] increased synovial PMNs of >80% [7] synovial CRP >6.9 mg/L

CONTACTS AND LOCATIONS:
Overall Officials: Ran Schwarzkopf, MD, Principal Investigator — NYU Langone
Locations (14):
- United States (14):
  - Eisenhower Health, Rancho Mirage, California
  - Centura Health, Denver, Colorado
  - Cleveland Clinic Florida, Weston, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - New England Baptist Hospital, Boston, Massachusetts
  - The Orthopedic Institute of New Jersey, Sparta, New Jersey
  - New York University Dept of Orthopedic Surgery, New York, New York
  - Hospital for Special Surgery, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Columbia, New York, New York
  - St. Francis Hospital, Roslyn, New York
  - Cleveland Clinic Ohio, Cleveland, Ohio